CLINICAL TRIAL: NCT02084511
Title: Effectiveness and Safety of Different Doses of BI 1026706 in Patients With Postoperative Dental Pain (a Single-centre, Partially Double-blinded, Randomised, placebo-and Active Comparator-controlled, Single-dose, Parallel-group Study)
Brief Title: Effectiveness and Safety of Different Doses of BI 1026706 in Patients With Postoperative Dental Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1320.13; 2013-003580-62 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib

ARMS (4):
- BI 1026706 low dose (Experimental): BI 1026706 low dose
  Interventions: Drug: Placebo to BI 1026706 solution; Drug: BI 1026706; Drug: Placebo to BI 1026706 tablet
- BI 1026706 high dose (Experimental): BI 1026706 high dose
  Interventions: Drug: BI 1026706; Drug: Placebo to BI 1026706 tablet
- Placebo reference (Experimental): Placebo reference
  Interventions: Drug: Placebo to BI 1026706 solution; Drug: Placebo to BI 1026706 tablet
- Celecoxib reference (Experimental): Celecoxib capsule
  Interventions: Drug: Placebo to BI 1026706 solution; Drug: Celecoxib

INTERVENTIONS:
Drug: Placebo to BI 1026706 solution — Placebo to BI 1026706 solution
  Arms: BI 1026706 low dose; Celecoxib reference; Placebo reference
Drug: BI 1026706 — BI 1026706
  Arms: BI 1026706 high dose; BI 1026706 low dose
Drug: Placebo to BI 1026706 tablet — Placebo to BI 1026706 tablet
  Arms: BI 1026706 high dose; BI 1026706 low dose; Placebo reference
Drug: Celecoxib — Celecoxib capsule
  Arms: Celecoxib reference

SUMMARY:
To investigate the effectiveness of BI 1026706 powder for reconstitution of an oral solution compared to placebo and the relative effectiveness compared to Celecoxib.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (Blood Pressure,Pulse Rate), 12-lead electrocardiogram, and clinical laboratory tests
2. Age 18 to 55 years (incl.)
3. Body Mass Index 18.5 to 29.9 kg/m2 (incl.)
4. Patients scheduled for removal of one mandibular third molar with partial or complete bony impaction. If medically indicated, the ipsilateral third molar in the upper jaw could also be removed;
5. Surgery will be conducted under local anaesthesia using 12% lidocaine (with epinephrine). Intravenous sedations and general anaesthetics are not permitted.
6. Reliable, cooperative, and of adequate intelligence to record the requested information on the analgesic questionnaire form
7. Examined by the attending oral surgeon or physician and medically cleared to participate in the study
8. Scheduled to undergo a qualifying surgical procedure
9. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including Blod Pressure, Pulse Rate or electrocardiogram) deviating from normal and judged clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged clinically relevant by the investigator
5. Acute local infection at the time of surgery that could confound the post-surgical evaluation
6. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
7. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1320.13.39001 Boehringer Ingelheim Investigational Site, Verona, Italy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, placebo and active comparator-controlled, partially double-blinded, single-dose, parallel-group, single-centre trial in male patients in double dummy design investigating 4 different treatments.
Groups:
- BI 50 mg PfOS: This trial has double dummy design, thus subjects were orally administered single dose of 50 mg of Boehringer Ingelheim (BI) 1026706 powder for oral solution (PfOS) with 200 mL of water plus matching placebo to BI 1026706 PfOS (to have 80 mL volume in total) and a placebo film-coated tablet.
- BI 200 mg PfOS: This trial has double dummy design, thus subjects were orally administered single dose of 200 mg of BI 1026706 powder for oral solution (PfOS) with 200 mL of water and a placebo film-coated tablet.
- Placebo: This trial has double dummy design, thus subjects were orally administered single dose of matching placebo to BI 1026706 powder for oral solution with 200 mL of water and placebo film coated tablet.
- Celecoxib 200 mg: This trial has double dummy design, thus subjects were orally administered single dose of Celecoxib hard capsule of 200 mg with 200 mL of water plus matching placebo to BI 1026706 PfOS.
Period: Overall Study
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: The treated set (TS) included all randomised patients who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.0 (8.7) | 24.2 (6.0) | 26.9 (5.7) | 26.5 (7.8) | 26.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: SPID0-8h
Description: Time-weighted sum of pain intensity difference (PID) from 0 to 8 hours post drug administration (SPID0-8h). SPID0-8h: possible range (-400; 800). The greater SPID0-8 the greater the reduction of pain intensity over the first 8 hours post drug administration.
Time Frame: up to 8 hours post drug administration
Population: The pharmacodynamic set (PD set) included all subjects of the Treated set (TS) who provided at least 1 primary or secondary PD endpoint value that was not flagged for exclusion.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on scale | -50.14 [-123.5 to 23.2] | -24.06 [-97.4 to 49.3] | -77.54 [-150.9 to -4.2] | 124.47 [51.1 to 197.8]
Statistical Analysis 1: Comparison: BI 50 mg PfOS vs Placebo; ANCOVA model was used with 'treatment' as fixed effect, 'patient baseline pain intensity (BPI)' as continuous covariate and the residual error term; Test type: Superiority or Other; Mean Difference (Final Values) = 27.39, 95% CI 2-sided [-76.3 to 131.1] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 2: Comparison: BI 200 mg PfOS vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 53.48, 95% CI 2-sided [-50.2 to 157.1] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 3: Comparison: BI 50 mg PfOS vs Celecoxib 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -174.61, 95% CI 2-sided [-278.3 to -70.9] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 4: Comparison: BI 200 mg PfOS vs Celecoxib 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -148.53, 95% CI 2-sided [-252.4 to -44.7] — Mean difference (final values) is actually the Least square mean

2. Secondary Outcome: TOTPAR0-8h
Description: Time-weighted total pain relief (PAR) from 0 to 8 hours (TOTPAR0-8h). (TOTPAR0-8h)TOTPAR0-8h: possible range (0;32). The greater TOTPAR0-8h the more pain relief was experienced over the first 8 hours post drug administration.
Time Frame: up to 8 hours post drug administration
Population: PD Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on scale | 3.85 [1.0 to 6.7] | 3.14 [0.3 to 6.0] | 2.16 [-0.7 to 5.0] | 10.12 [7.3 to 13.0]
Statistical Analysis 1: Comparison: BI 50 mg PfOS vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.70, 95% CI 2-sided [-2.3 to 5.7] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 2: Comparison: BI 200 mg PfOS vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Median Difference (Final Values) = 0.98, 95% CI 2-sided [-3.0 to 5.0] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 3: Comparison: BI 50 mg PfOS vs Celecoxib 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -6.27, 95% CI 2-sided [-10.3 to -2.2] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 4: Comparison: BI 200 mg PfOS vs Celecoxib 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -6.98, 95% CI 2-sided [-11.0 to -2.9] — Mean difference (final values) is actually the Least square mean

3. Secondary Outcome: SPID0-2h
Description: Time-weighted sum of PID from 0 to 2 hours (SPID0-2h). SPID0-2h: possible range (-100; 200). The greater SPID0-2 the greater the reduction of pain intensity over the first 2 hours post drug administration.
Time Frame: up to 2 hours post drug administration
Population: PD set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on scale | -8.08 [-23.6 to 7.4] | 6.57 [-8.9 to 22.1] | -14.01 [-29.5 to 1.5] | 5.20 [-10.3 to 20.7]
Statistical Analysis 1: Comparison: BI 50 mg PfOS vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 5.93, 95% CI 2-sided [-16.0 to 27.8] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 2: Comparison: BI 200 mg PfOS vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 20.58, 95% CI 2-sided [-1.3 to 42.5] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 3: Comparison: BI 50 mg PfOS vs Celecoxib 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -13.29, 95% CI 2-sided [-35.2 to 8.6] — Mean difference (final values) is actually the Least square mean
Statistical Analysis 4: Comparison: BI 200 mg PfOS vs Celecoxib 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [-20.6 to 23.3] — Mean difference (final values) is actually the Least square mean

4. Secondary Outcome: Time to Meaningful Pain Relief
Description: Time to meaningful pain relief was captured by a stopwatch started by the trial staff immediately after administration of study medication and stopped by the subject as soon as a meaningful pain relief was felt by the subject. If a subject did not have any meaningful pain relief up to 10 h, the time was censored at 10 h.
  Kaplan-Meier estimates over time for each treatment and time to event endpoint 'Time to meaningful pain relief' were presented descriptively.
Time Frame: up to 10 hours post drug administration
Population: PD set
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
hours | 5.00 [NA to NA] — Due to low number of events, 95% Confidence interval was not estimable thus not reported. | 2.67 [2.67 to NA] — Due to low number of events, Upper limit of the 95% Confidence interval was not estimable thus not reported. | NA [NA to NA] — Due to only one event reported, Median and 95% Confidence interval was not estimable thus not reported. | 1.93 [1.25 to 2.37]
Statistical Analysis 1: Comparison: BI 50 mg PfOS vs Placebo; Log rank test used to evaluate the difference between each active treatment and placebo; Test type: Superiority or Other; p = 0.2503, Log Rank
Statistical Analysis 2: Comparison: BI 200 mg PfOS vs Placebo; Log rank test used to evaluate the difference between each active treatment and placebo; Test type: Superiority or Other; p = 0.1851, Log Rank
Statistical Analysis 3: Comparison: Placebo vs Celecoxib 200 mg; Log rank test used to evaluate the difference between each active treatment and placebo; Test type: Superiority or Other; p = 0.0167, Log Rank

5. Secondary Outcome: Time to First Dose of Rescue Medication
Description: The time to first dose of rescue medication was defined by the difference in time of the study drug intake and the time of first rescue medication use within the first 10 h after study drug administration.
  Kaplan-Meier estimates over time for each treatment and time to event endpoint 'Time to first dose of rescue medication' were presented descriptively.
  Subjects without intake of rescue medication within the first 10 hours after study drug administration were censored at 10 hours.
Time Frame: up to 10 hours post drug administration
Population: PD set
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
hours | 1.57 [1.10 to 2.27] | 1.53 [1.35 to 2.08] | 1.52 [1.17 to 1.58] | NA [1.25 to NA] — Due to low number of events, median and upper limit of the 95% Confidence interval was not estimable.
Statistical Analysis 1: Comparison: BI 50 mg PfOS vs Placebo; Log rank test used to evaluate the difference between each active treatment and placebo; Test type: Superiority or Other; p = 0.4150, Log Rank
Statistical Analysis 2: Comparison: BI 200 mg PfOS vs Placebo; Log rank test used to evaluate the difference between each active treatment and placebo; Test type: Superiority or Other; p = 0.3093, Log Rank
Statistical Analysis 3: Comparison: Placebo vs Celecoxib 200 mg; Log rank test used to evaluate the difference between each active treatment and placebo; Test type: Superiority or Other; p = 0.0074, Log Rank

6. Secondary Outcome: Percentage of Patients With Drug-related Adverse Events
Description: Percentage of patients with drug-related adverse events
Time Frame: From first drug administration until 3 days after last drug administration, upto 4 days
Population: Treated Set
Measure: Number; unit: Percentage of participants
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 days after last drug administration, upto 4 days
Arm/Group | BI 50 mg PfOS | BI 200 mg PfOS | Placebo | Celecoxib 200 mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.